CLINICAL TRIAL: NCT04893824
Title: Grappler® Interference Screw Post-Market Clinical Follow-Up Study
Status: Completed | Type: Observational
Sponsor: Paragon 28 (Industry)
Responsible Party: Sponsor
Other Study IDs: P41-SP-0001
Record Dates: First submitted 2021-05-11; First posted 2021-05-20 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2022-03

CONDITIONS: Ankle Injuries; Syndesmotic Injuries; Ankle Inversion Sprain; Deltoid Ankle Sprain; Achilles Tendon Rupture; Flexor Hallucis Longus on the Left; Flexor Digitorum Longus on the Left; Ankle Sprains; Flexor Hallucis Longus on the Right; Flexor Digitorum Longus on the Right
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Grappler® Interference Screw System — Foot and/or ankle procedure involving soft tissue attachment to bone using the Grappler® Interference Screw System

SUMMARY:
Ambispective, multi-surgeon, single site, consecutive case series to determine the safety, performance, and benefits of the Grappler(R) Interference Screw.

DETAILED DESCRIPTION:
This is a ambispective, multi-surgeon, single site, consecutive case series. Data collection will occur in two phases. Retrospective data collection will occur upon subject identification, and data will be collected from the site's medical records for minimum of 50 subjects who have undergone soft tissue to bone fixation with the Grappler® Interference Screw System. Data will be collected from the subjects' pre-op visits, intra-op visits, 7 week post-op follow-up visits (± 4 weeks), and 6 month post-op follow-up visits (± 4 weeks). The subject must have adequate radiographic and medical records for the minimum follow up requirement of 6 months. Prospective data collection will occur upon subject's provision of written informed consent, and data will be collected from patient reported outcomes (PRO's).

ELIGIBILITY:
Inclusion Criteria:

* The subject must have undergone a foot and/or ankle procedure involving soft tissue attachment to bone using the Grappler® Interference Screw System and completed by one of the designated investigators who are experienced in the use of such implants and the required specialized surgical techniques
* The subject must have adequate radiographic and medical records for the minimum follow-up requirement of six months

For the Prospective Data Collection:

- The subject is willing to provide written informed consent

Exclusion Criteria:

* None

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The investigational population will include a minimum of 50 subjects who have undergone a foot and/or ankle procedure that fulfill the eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2022-03-11 (Actual); Study Completion 2022-03-25 (Actual)

PRIMARY OUTCOMES:
Incidence of revisions | 6 Months Post-Op
  Safety will be assessed by recording the incidence of revisions. The relationship of events will be attributed to either the implant or instrumentation.
Incidence of adverse events | 6 Months Post-Op
  Safety will be assessed by recording the incidence of adverse events. The relationship of events will be attributed to either the implant or instrumentation.
Incidence of complications | 6 Months Post-Op
  Safety will be assessed by recording the incidence of complications. The relationship of events will be attributed to either the implant or instrumentation.

SECONDARY OUTCOMES:
Rate of recurrence of deformity | 7 Weeks Post-Op, 6 Months Post-Op
  Safety as related to rate of recurrence of deformity
Rate of implant failure | Intra-Op, 7 Weeks Post-Op, 6 Months Post-Op
  Safety as related to rate of implant failure
Rate of re-tear or re-rupture of fixated soft tissue | 7 Weeks Post-Op, 6 Months Post-Op
  Safety as related to rate of re-tear or re-rupture of fixated soft tissue
Rate of screw removal | 7 Weeks Post-Op, 6 Months Post-Op
  Safety as related to rate of screw removal
Foot and Ankle Mobility Measure | 6 months post-operative
  Device performance and benefits as related to Foot and Ankle Mobility Measure Activities of Daily Living (0-84) and sports (0-32) subscales. The higher the score, the higher the level of function, with 100% representing no dysfunction.
Visual Analog Scale | 6 months post-operative
  Device performance and benefits as related to pain levels based on the Visual Analog Scale (range: 0 to 100; 0 = no pain; 100 = worst pain imaginable)
Patient satisfaction | 6 months post-operative
  Device performance and benefits as related to patient satisfaction (very satisfied, good, fair, not satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Jacy Legue, Study Director — Paragon 28
Locations (1):
- Orthopedic Foot and Ankle, Worthington, Ohio, United States

IPD SHARING:
Plan to Share IPD: No